CLINICAL TRIAL: NCT05659498
Title: Cardiac Rehabilitation for Cardiovascular Risk Reduction in People With Severe and Persistent Mental Illness: A Pilot Randomized Study
Brief Title: Cardiac Rehabilitation for Cardiovascular Risk Reduction in People With Severe and Persistent Mental Illness
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Lady Davis Institute (Other)
Collaborators: Jewish General Hospital (Other)
Responsible Party: Principal Investigator, Michael Goldfarb, Attending Staff, Division of Cardiology, Lady Davis Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 20233395
Record Dates: First submitted 2022-12-05; First posted 2022-12-21 (Actual); Last update posted 2023-03-10 (Actual); Status verified 2023-03

CONDITIONS: Mental Illness Persistent; Cardiovascular Prevention
Keywords: Severe and persistent mental illness; Primary prevention; Measures; Schizophrenia; Schizoaffective disorder; Bipolar disorder
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Bipolar Disorder

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Masking the participant and provider is not possible due to the nature of the intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The standard cardiac rehabilitation program consists of the following: a (1) consultation with a kinesiologist to assess level of fitness and to prepare an individually customized exercise plan, (2) consultation with a dietitian to guide the participant with healthy nutrition choices, (3) on site supervised and/or virtual exercise sessions with gradual elaboration of a home program, (4) weekly educational capsules and monthly workshops related to cardiac health, and, (5) if deemed necessary by the treating team, consultation with a psychologist, an occupational therapist, a physiotherapist, or a social worker.
  Interventions: Behavioral: Cardiac Rehabilitation Program
- Control (No Intervention): Participants in the control group will receive educational information on maintaining optimal cardiovascular health. Participants will be encouraged to undergo 30 minutes of moderate-intensity aerobic activity at least 5 days per week. Participants will be given educational materials on recommended diet and exercise.

INTERVENTIONS:
Behavioral: Cardiac Rehabilitation Program — The standard cardiac rehabilitation program consists of the following: a (1) consultation with a kinesiologist to assess level of fitness and to prepare an individually customized exercise plan, (2) consultation with a dietitian to guide the participant with healthy nutrition choices, (3) on site supervised and/or virtual exercise sessions with gradual elaboration of a home program, (4) weekly educational capsules and monthly workshops related to cardiac health, and, (5) if deemed necessary by the treating team, consultation with a psychologist, an occupational therapist, a physiotherapist, or a social worker.
  Arms: Intervention

SUMMARY:
The goal of this prospective, randomized trial is to explore the link between cardiovascular disease and mortality in individuals with severe and persistent mental illness (SPMI). The main question it aims to answer is: Is a primary prevention cardiac rehabilitation intervention feasible and effective at reducing cardiovascular risk in people with a primary psychotic disorder or bipolar disorder?"

Participants will undergo a multi-component primary prevention intervention program. Researchers will compare with a control group to see if cardiovascular risk reduction is attained.

DETAILED DESCRIPTION:
This prospective, randomized study aims to recruit 46 adults with schizophrenia, schizoaffective disorder, or bipolar disorder, who are classified as intermediate or high 10-year risk for a cardiovascular event, into a multi-component cardiac rehabilitation intervention program. The aim is to explore the feasibility and efficacy of this multi-component primary prevention intervention program in reducing cardiovascular risk in individuals with SPMI.

Evidence supports a high burden of cardiovascular disease and mortality in individuals with SPMI. In link, multiple studies outline disparities in access to quality cardiovascular care in people with SPMI. Given the high CV risk factor burden in people with SPMI and the disparity in access and quality of care, there is a need to screen for CV risk factors and initiate and monitor guideline-directed therapies in people with SPMI.

Intervention outcomes will be measured using the Framingham 10-year cardiovascular risk score, the Framingham 30-year cardiovascular risk score, the PRIMOSE BMI and Lipid risk scores, the EQ-5D-5L scale and the CGI score. Continuous variables will be displayed as means, with associated standard deviations. Categorical variables will be represented as frequencies and percentages. Subsequent comparative analysis will take place, where the overall cohort will be characterized into high risk (top quartile) and low risk (bottom quartile) cohorts. This will be accomplished using the chi-squared test or the Fisher exact test, along with the student's t test and the Mann-Whitney U test when appropriate. SPSS 24.0 will be the statistical software used.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 30 to 59 years old
* Psychiatric diagnosis of schizophrenia, schizoaffective disorder, or bipolar I disorder
* 2 or more cardiac risk behaviors or conditions: smoking, obese, hypertension, diabetes, metabolic syndrome, dyslipidemia, obstructive sleep apnea
* 10-year Framingham cardiovascular risk score of ≥ 10% (intermediate risk)
* Willing to participate in cardiac rehabilitation program

Exclusion Criteria:

* Psychiatric instability, as judged by treating psychiatrist
* Distance from cardiac rehabilitation centre that would preclude participation
* Unsafe to participate in the cardiac rehabilitation intervention, as judged by the cardiology assessment
* Pregnant
* Known coronary artery disease, cerebrovascular disease, or peripheral vascular disease
* Court ordered mandatory or tutor

Ages: 30 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Estimated)
Dates: Start 2022-12-14 (Actual); Primary Completion 2024-05 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
Efficacy outcome | 9 months
  10-year Framingham cardiovascular risk score

SECONDARY OUTCOMES:
30-year Cardiovascular risk | 9 months
  30-year Framingham cardiovascular risk score
PRIMROSE BMI risk score | 9 months
  PRIMROSE BMI risk score
PRIMROSE Lipid risk score | 9 months
  PRIMROSE Lipid risk score
Quality of life | 9 months
  EQ-5D-5L

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Goldfarb, Principal Investigator — Lady Davis Institute
Locations (1):
- Jewish General Hospital/Lady Davis Institute, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Daumit GL, Dalcin AT, Dickerson FB, Miller ER, Evins AE, Cather C, Jerome GJ, Young DR, Charleston JB, Gennusa JV 3rd, Goldsholl S, Cook C, Heller A, McGinty EE, Crum RM, Appel LJ, Wang NY. Effect of a Comprehensive Cardiovascular Risk Reduction Intervention in Persons With Serious Mental Illness: A Randomized Clinical Trial. JAMA Netw Open. 2020 Jun 1;3(6):e207247. doi: 10.1001/jamanetworkopen.2020.7247. PMID 32530472
- [Background] Nielsen RE, Banner J, Jensen SE. Cardiovascular disease in patients with severe mental illness. Nat Rev Cardiol. 2021 Feb;18(2):136-145. doi: 10.1038/s41569-020-00463-7. Epub 2020 Oct 30. PMID 33128044
- [Background] Goldfarb M, De Hert M, Detraux J, Di Palo K, Munir H, Music S, Pina I, Ringen PA. Severe Mental Illness and Cardiovascular Disease: JACC State-of-the-Art Review. J Am Coll Cardiol. 2022 Aug 30;80(9):918-933. doi: 10.1016/j.jacc.2022.06.017. PMID 36007991